CLINICAL TRIAL: NCT01611051
Title: A Study Comparing Pegylated rhG-CSF and rhG-CSF as Support to Breast Cancer Patients Receiving Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HHPG-19K -III-01
Record Dates: First submitted 2012-05-31; First posted 2012-06-04 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2013-01

CONDITIONS: Breast Cancer; Neutropenia; Febrile Neutropenia
Keywords: breast cancer; neutropenia; febrile neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia; Febrile Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pegylated rhG-CSF: 100µg/kg (Experimental): Chemtherapy naive patients receiving chemotherapy and Pegylated rhG-CSF 100µg/kg
  Interventions: Drug: Drug: Pegylated rhG-CSF: 100µg/kg
- Pegylated rhG-CSF: 6mg (Experimental): Chemtherapy naive patients receiving chemotherapy and Pegylated rhG-CSF 6mg
  Interventions: Drug: Pegylated rhG-CSF: 6mg
- rhG-CSF 5ug/kg/day (Active Comparator): Chemtherapy naive patients receiving chemotherapy and rhG-CSF 5ug/kg/day
  Interventions: Drug: rhG-CSF 5ug/kg/day

INTERVENTIONS:
Drug: Drug: Pegylated rhG-CSF: 100µg/kg — Patients were administered pegylated rhG-CSF 100 ug/kg once at the 3rd day of every chemotherapy cycle. Chemotherapy regimen: EC (epirubicin 100 mg/m2 +cyclophosphamide 600 mg/m2) or ET (epirubicin 75 mg/m2 + docetaxel 75 mg/m2).
  Arms: Pegylated rhG-CSF: 100µg/kg
Drug: Pegylated rhG-CSF: 6mg — Patients were administered pegylated rhG-CSF 6mg once at the 3rd day of every chemotherapy cycle. Chemotherapy regimen: EC (epirubicin 100 mg/m2 +cyclophosphamide 600 mg/m2) or ET (epirubicin 75 mg/m2 + docetaxel 75 mg/m2).
  Arms: Pegylated rhG-CSF: 6mg
Drug: rhG-CSF 5ug/kg/day — Patients were administered pegylated rhG-CSF 6 ug/kg/day from the 3rd day of every chemotherapy cycle. Chemotherapy regimen: EC (epirubicin 100 mg/m2 +cyclophosphamide 600 mg/m2) or ET (epirubicin 75 mg/m2 + docetaxel 75 mg/m2).
  Arms: rhG-CSF 5ug/kg/day

SUMMARY:
Neutropenia is one of the most frequent adverse effects of chemotherapy, and the main factor to limit the dosage and the continuation of chemotherapy. A newly pegylated rhG-CSF was independently developed by JIANGSU HENGRUI Medicine Co., Ltd, China. Phase 1a, 1b and phase 2 trials have shown that pegylated rhG-CSF has decreased renal clearance, increased plasma half-life, and prolonged efficacy in compare with rhG-CSF. The purpose of this study is to determine the safety and effectiveness of pegylated rhG-CSF in preventing neutropenia following chemotherapy in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Investigator diagnosis of breast cancer
* Age 18 to 70 years
* ECOG performance status ≤ 1
* Chemotherapy naïve
* Body weight ≥ 45kg
* Hemoglobin ≥ 90g/L; white blood cell ≥ 4.0×109/L; absolute neutrophil count ≥1.5 × 109/L; platelet count ≥ 100 × 109/L
* Alanine transarninase ≤1.5×ULN; aspartate aminotransferase ≤1.5×ULN; serum creatinine ≤1.5×ULN; total bilirubin ≤1.5×ULN

Exclusion Criteria:

* Prior bone marrow or stem cell transplantation
* Received systemic antibiotics treatment within 72 h of chemotherapy
* Radiation therapy within 4 weeks of randomization into this study
* Pregnancy, lactation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Rate and the duration of grade 3/4 neutropenia in cycle 1 | 21 days
  Proportion and the duration of subjects developing ANC lower than 1.0 × 109/L.

SECONDARY OUTCOMES:
Rate and the duration of grade 3/4 neutropenia in cycle 2-4 | Through cycle 2 to cycle 4
  Proportion and the duration of subjects developing ANC lower than 1.0 × 109/L from cycle 2 to cycle 4.
Rate of the febrile neutropenia in cycle 1 | Through 4 cycles
  Rate of ANC<0.5×109/L and auxiliary temperature>38.5℃.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Affiliated to Academy Military Medical Science, Beijing, Beijing Municipality, China